CLINICAL TRIAL: NCT03064048
Title: Effect of Nitric Oxide (NO) Supplementation on Neurocognitive Measures in Argininosuccinate Lyase Deficiency (ASLD)
Brief Title: Nitric Oxide Supplementation on Neurocognitive Functions in Patients With ASLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); Neogenis Laboratories (Other)
Responsible Party: Principal Investigator, Sandesh Chakravarthy Sreenath Nagamani, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-40143
Record Dates: First submitted 2017-02-10; First posted 2017-02-24 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Argininosuccinate Lyase Deficiency; Urea Cycle Disorder; Urea Cycle Disorders, Inborn; Argininosuccinic Aciduria
Keywords: Argininosuccinate Lyase Deficiency; Urea Cycle Disorder
MeSH Terms: conditions — Argininosuccinic Aciduria; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Intervention Model Description: Active Comparator: Nitric oxide supplement Active Comparator will l not contain nitric oxide supplement.
  Placebo Comparator: Placebo Placebo will not contain nitric oxide supplement.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization for treatment assignment is by the providing Institution's Investigational Pharmacy Services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neo-ASA (Active Comparator): During this arm the participant will receive a lozenge with nitric oxide as a dietary supplement twice daily.
  Interventions: Dietary Supplement: Neo-ASA
- Placebo (Placebo Comparator): During this arm the participant will receive a lozenge which will not contain nitric oxide as a dietary supplement twice daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Neo-ASA — Dietary supplement with nitric oxide in the form of a lozenge called Neo-ASA.
  Arms: Neo-ASA
Dietary Supplement: Placebo — Dietary supplement with no nitric oxide in the form of a lozenge to look and taste like the dietary supplement Neo-ASA
  Arms: Placebo

SUMMARY:
This is a study involving a dietary supplement. Patients with argininosuccinate lyase deficiency (ASLD) will be randomly assigned to receive either a nitric oxide dietary supplement or placebo for 24 weeks, and then crossed-over to receive the other treatment for 24 weeks. The investigators will assess the effects of the supplement in domains of general cognition, memory, executive functioning, and fine motor functioning in individuals with ASLD.

DETAILED DESCRIPTION:
Argininosuccinate lyase deficiency (ASLD; also known as argininosuccinic aciduria) is the second most common urea cycle disorder (UCD) and accounts for 15-20% of all disorders of ureagenesis. Individuals with ASLD can have unique clinical and physiologic characteristics as compared to other UCDs. Previous work from the members of the UCDC have shown that in spite of having fewer episodes of hyperammonemia as compared to those with proximal blockade of the urea cycle, individuals with ASLD can develop intellectual and learning disabilities. Neurocognitive deficits have been observed even in individuals without any documented hyperammonemia. Furthermore, hepatic abnormalities including hepatomegaly, hepatic injury, fibrosis and even frank cirrhosis, and vascular issues like hypertension are well known in the disorder. Previous work from the members of the UCDC has demonstrated a tissue- and molecular-specific role for ASL in the generation of NO. ASL is not only required for the synthesis of L-arginine, the substrate for the synthesis of NO, but is also an integral member of a complex that is critical for synthesis of NO from arginine. Loss of ASL can thus lead to systemic and tissue-specific NO deficiencies, which could potentially contribute to the complex phenotype including the neurocognitive deficits. A rational therapeutic option would hence be to use a NOS-independent NO supplement.

The purpose of this study is to determine whether a dietary NO supplement, Neo-ASA, would improve general cognition, memory, executive functioning, fine motor functioning, and attention in individuals with ASLD. In this single-center trial, double-blind, randomized, placebo-controlled, crossover study, individuals with ASLD will be assigned to receive a medication containing NO dietary supplement for 24 weeks and a placebo for 24 weeks. General cognition, memory, executive functioning, and fine motor functioning will be assessed and compared at the end of treatment with placebo and Neo-ASA.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 6 and <50 years
2. Diagnosis of ASLD confirmed by biochemical OR enzymatic OR genetic testing
3. Has a history of compliance with diet and treatment
4. Negative pregnancy test and ability to use birth control method for the entire duration of the study (if the subject is of child-bearing potential)
5. Males who enroll in the study (and their partners) should argee to use an acceptable form of birth control for the entire duration of the study

Exclusion Criteria:

1. Clinical or laboratory abnormality of Grade 3 or greater according to the CTCAE (or for conditions not covered by the CTCAE, a severe or life-threatening toxicity) at enrollment which, in the view of the investigator compromises safety. (Elevated plasma levels of aspartate and alanine aminotransferases, or low serum potassium will not be considered as exclusion criteria as these are phenotypic manifestations of ASLD.)
2. Known hypersensitivity to Neo-ASA or nitrite
3. Individuals currently being administered other investigational agents

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Delis-Kaplan Executive Function System - Tower subtest | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Stanford-Binet - 4th Edition: Bead Memory and Sentence Memory subtests | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Grip Strength | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Grooved Pegboard | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Wechsler Intelligence Scale for Children OR Wechsler Adult Intelligence Scale - 4th Edition (in subjects > 16 years of age) | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Tower of London Test | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo
Conners Continuous Performance Test - 3rd Edition Conners Continuous Performance Test - 3rd Edition | 24 weeks
  Change in the scores from baseline to 24 weeks with drug vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sandesh C Nagamani, M.D., Principal Investigator — Baylor College of Medicine; Brendan Lee, M.D., PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the policy of the National Institutes of Health (one of the study sponsors) research data may be put in a secure, limited-access database known as dbGaP. The data will include any genetic test results as well as other information about medical problems. There will be NO identifiers included (no name, data of birth, address, social security number, etc.). Access to this information is restricted by the National Institutes of Health. Only doctors and scientists who get approval from the National Institutes of Health can access this de-identified data.

REFERENCES:
- [Background] Nagamani SC, Campeau PM, Shchelochkov OA, Premkumar MH, Guse K, Brunetti-Pierri N, Chen Y, Sun Q, Tang Y, Palmer D, Reddy AK, Li L, Slesnick TC, Feig DI, Caudle S, Harrison D, Salviati L, Marini JC, Bryan NS, Erez A, Lee B. Nitric-oxide supplementation for treatment of long-term complications in argininosuccinic aciduria. Am J Hum Genet. 2012 May 4;90(5):836-46. doi: 10.1016/j.ajhg.2012.03.018. Epub 2012 Apr 26. PMID 22541557
- [Background] Nagamani SCS, Burrage LC, Lee B. Argininosuccinate Lyase Deficiency. 2011 Feb 3 [updated 2025 Aug 14]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK51784/ PMID 21290785
- [Background] Erez A, Nagamani SC, Shchelochkov OA, Premkumar MH, Campeau PM, Chen Y, Garg HK, Li L, Mian A, Bertin TK, Black JO, Zeng H, Tang Y, Reddy AK, Summar M, O'Brien WE, Harrison DG, Mitch WE, Marini JC, Aschner JL, Bryan NS, Lee B. Requirement of argininosuccinate lyase for systemic nitric oxide production. Nat Med. 2011 Nov 13;17(12):1619-26. doi: 10.1038/nm.2544. PMID 22081021